CLINICAL TRIAL: NCT04417335
Title: Reducing Hospital Admission of Elderly in SARS-CoV-2 Pandemic Via the Induction of Trained Immunity by Bacillus Calmette-Guérin Vaccination, a Randomized Controlled Trial
Brief Title: Reducing COVID-19 Related Hospital Admission in Elderly by BCG Vaccination
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL73430.091.20; 2020-001591-15 (EudraCT Number)
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: BCG; Bacille Calmette-Guérin; COVID-19; SARS-CoV-2; trained immunity; off-target effects
MeSH Terms: conditions — COVID-19 | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: placebo-controlled adaptive multi-centre randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): BCG vaccine (Danish strain 1331, SSI, Denmark)
  Interventions: Biological: BCG vaccine
- Placebo (Placebo Comparator): 0.9% NaCl
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BCG vaccine — Bacille Calmette-Guérin is a live attenuated strain of Mycobacterium bovis developed in 1921 to prevent tuberculosis and other mycobacterial related infections.
  Arms: Treatment
Biological: Placebo — 0.9% NaCl
  Arms: Placebo

SUMMARY:
Bacillus Calmette-Guérin (BCG) vaccine not only protects against tuberculosis, but has also been shown to induce protection against various infections with a viral aetiology, leading to significant reductions in morbidity and mortality. We hypothesize that BCG vaccination might be a potent preventive measure against SARS-CoV-2 infection and/or may reduce disease severity in elderly people, who are known to be at increased risk of illness and death from SARS-CoV-2 infection.

Therefore, we will in this placebo-controlled adaptive multi-centre randomized controlled trial evaluate the ability of BCG to reduce hospital admission and its efficacy to improve the clinical course of SARS-CoV-2 infection in elderly people((≥ 60 years of age).

DETAILED DESCRIPTION:
On March 11 2020 the World Health Organization (WHO) declared the coronavirus (SARS-CoV-2) outbreak a pandemic. The number of confirmed cases continues to rise, leading to significant morbidity and mortality worldwide. Although individuals of any age can acquire SARS-CoV-2, adults of middle age and older are most commonly affected. Moreover, recent reports demonstrate that mortality rates rise significantly among patients 60 years and older. Therefore, strategies to prevent SARS-CoV-2 infection or to reduce its clinical consequences in elderly are desperately needed. Bacillus Calmette-Guérin (BCG) vaccine not only protects against tuberculosis, but has also been shown to induce protection against various infections with a viral aetiology, leading to significant reductions in morbidity and mortality. We hypothesize that BCG vaccination may reduce hospital admission and improve the clinical course of symptoms of elderly people during the SARS-CoV-2 outbreak. Primary objective: To reduce hospital admission of community dwelling older persons during the pandemic of SARS-CoV-2. Secondary objective: To reduce disease severity, the duration of hospital admission, ICU admission, or death in elderly during the pandemic of SARS-CoV-2.

Study design: A placebo-controlled adaptive multi-centre randomized controlled trial.

Study population: Elderly people (≥ 60 years of age). Intervention: Participants will be randomized between intracutaneous administration of BCG vaccine or placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 60 years)

Exclusion Criteria:

* Fever (>38 ºC) within the past 24 hours
* Suspicion of current active viral or bacterial infection
* Expected vaccination during the first three months of the study period
* Severely immunocompromised subjects. This exclusion category comprises: a) subjects with known infection by the human immunodeficiency virus (HIV-1); b) neutropenic subjects with less than 500 neutrophils/mm3; c) subjects with solid organ transplantation; d) subjects with bone marrow transplantation; e) subjects under chemotherapy; f) subjects with primary immunodeficiency; g) severe lymphopenia with less than 400 lymphocytes/mm3; h) treatment with any immunosuppressant drugs such as anti-cytokine therapies, and treatment with oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than 3 months, or probable use of oral or intravenous steroids in the following four weeks.
* Active solid or non-solid malignancy or lymphoma within the prior two years
* Active participation in another research study that involves BCG administration

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2014 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 related hospital admission | Maximum of 1 year

SECONDARY OUTCOMES:
the duration of hospital admission due to documented COVID-19 | Maximum of 1 year
the cumulative incidence of documented SARS-CoV-2 infection | Maximum of 1 year
the cumulative incidence of self-reported acute respiratory symptoms or fever | Maximum of 1 year
the cumulative incidence of death due to documented SARS-CoV-2 infection | 1 year
the cumulative incidence of hospital admission for any reason | Maximum of 1 year
the cumulative incidence of Intensive Care Admission due to documented SARS-CoV-2 infection | Maximum of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboud University, Nijmegen, Gelderland
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fohse K, Taks EJM, Moorlag SJCFM, Bonten MJM, van Crevel R, Ten Oever J, van Werkhoven CH, Netea MG, van de Maat JS, Hoogerwerf JJ. The impact of circadian rhythm on Bacillus Calmette-Guerin vaccination effects on SARS-CoV-2 infections. Front Immunol. 2023 Feb 16;14:980711. doi: 10.3389/fimmu.2023.980711. eCollection 2023. PMID 36875134
- [Derived] Moorlag SJCFM, Taks E, Ten Doesschate T, van der Vaart TW, Janssen AB, Muller L, Ostermann P, Dijkstra H, Lemmers H, Simonetti E, Mazur M, Schaal H, Ter Heine R, van de Veerdonk FL, Bleeker-Rovers CP, van Crevel R, Ten Oever J, de Jonge MI, Bonten MJ, van Werkhoven CH, Netea MG. Efficacy of BCG Vaccination Against Respiratory Tract Infections in Older Adults During the Coronavirus Disease 2019 Pandemic. Clin Infect Dis. 2022 Aug 24;75(1):e938-e946. doi: 10.1093/cid/ciac182. PMID 35247264